CLINICAL TRIAL: NCT00630162
Title: Survey of Intestinal Protozoal Infections and Sexual Transmitted Diseases Among Targeted Cohorts
Brief Title: Intestinal Protozoal Infections and Sexual Transmitted Diseases Among Targeted Cohorts
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Other Study IDs: QM094008
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections; Protozoan Infections
Keywords: protozoa; Amoeba
MeSH Terms: conditions — HIV Infections; Protozoan Infections | interventions — S29X protein, Amoeba proteus symbiotic bacterium

INTERVENTIONS:
Genetic: amoeba

SUMMARY:
In this two-year study, we will target two high risk groups, including MSM of HIV-infected and those of non-HIV-infected. We will avail the serodiagnosis to detect the potential amebic carriers in both groups; and use microscopy to detect protozoas other than amebiasis. Meanwhile we will also survey the patients' status of sexual transmitted diseases (STD). For the amebic carriers, we will apply specific antigen and molecular biologic method to follow up the duration of the persistence of fecal amebas. We try to clarify the dynamic change of amebic carriage.

DETAILED DESCRIPTION:
HIV-infected persons who are men having sex with men (MSM) are prone to acquire invasive amebiasis. It would cast great threat for public health if the pathogens are spread by way of human to human transmission and food contamination.

From 2000 to 2004, we assessed the seroprevalence of Entamoeba histolytica infection using indirect hemagglutination antibody (IHA) assay among 667 HIV-infected persons (group 1), 1311 asymptomatic HIV-uninfected persons seeking anonymous HIV testing (group 2), 616 HIV-uninfected controls with gastrointestinal symptoms (diarrhea and/or liver abscess) seeking medical care (group 3), and 2500 healthy controls undergoing health check-up (group 4). An IHA titer greater than 128 was detected in 7.1% of group 1, 2.5% of group 2, 1.8% of group 3, and 0.1% of group 4 (p<0.0001). The highest seroprevalence (11.2%) was noted among HIV-infected persons who were MSM aged 30 to 39 years. Compared with persons with gastrointestinal symptoms, the adjusted odds ratio for having high IHA titers among HIV-infected persons was 3.206 (95% confidence interval, 1.433, 7.176) (p=0.005). These findings demonstrate that HIV-infected persons, especially MSM aged 30 to 39 years, are at significantly higher risk of E. histolytica infection.

In this two-year study, we will target two high risk groups, including MSM of HIV-infected and those of non-HIV-infected. We will avail the serodiagnosis to detect the potential amebic carriers in both groups; and use microscopy to detect protozoas other than amebiasis. Meanwhile we will also survey the patients' status of sexual transmitted diseases (STD). For the amebic carriers, we will apply specific antigen and molecular biologic method to follow up the duration of the persistence of fecal amebas. We try to clarify the dynamic change of amebic carriage.

We anticipate this study could outline the epidemiology and risk factors of protozoal infections and STD in MSM cohorts. We also hope to reduce the the infection rate (protozoa and HIV) and disease rate (STD) through the repetitively effective health education and consultation during the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV-1 Disease
* Clinical diagnosis of Intestinal protozoal infections

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-03; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, MD, Study Director — Chung-Ho Memorial Hospital,Kaohsiung Medical University
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshiung, Taiwan